CLINICAL TRIAL: NCT01502215
Title: Transfusion Requirements in Surgical Oncologic Patient
Acronym: TRISOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliano P Almeida, MD, Principal Investigator, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 002/11
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Red Blood Cells Transfusion; Oncologic Surgery
MeSH Terms: interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Liberal Transfusion Strategy (Active Comparator): Liberal Group - transfusion when hemoglobin is lower than 9 g/dL. Intervention: Other: Red blood cell transfusion
  Interventions: Other: Red blood cell transfusion
- Restrictive Transfusion Strategy (Active Comparator): Restrictive Group - transfusion when hemoglobin is lower than 7 g/dL Intervention: Other: Red blood cell transfusion
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — Red blood cell (RBC) transfusion will be given when hemoglobin fall below 9 g/dL since ICU admission until the discharge of intensive care unit. Following administration of the 1 RBC unit, a repeat hemoglobin levels is performed;if a patient's hemoglobin is 9 g/dL or higher, no additional transfusion is necessary.
  Arms: Liberal Transfusion Strategy
Other: Red blood cell transfusion — Red blood cell (RBC) transfusion will be only given when hemoglobin fall below 7 g/dL since ICU admission until the discharge of intensive care unit. Following administration of the 1 RBC unit, a repeat hematocrit is performed;if a patient's hemoglobin 7 g/dL or higher, no additional transfusion is necessary
  Arms: Restrictive Transfusion Strategy

SUMMARY:
Blood transfusion during perioperative period in patients undergoing to major surgery has been associated to several postoperative complications. Particularly in oncologic surgery, red blood cell transfusion has been investigated as a factor of worse outcome and cancer recurrence due to postoperative impairment of cellular immunity. Although red blood cell transfusion has decreased in worldwide clinical practice, this issue still remains a matter of controversy in oncologic surgery. There are no prospective studies comparing outcomes between restrictive or liberal of blood transfusion strategy in oncologic surgery. This study is a prospective and randomized study comparing clinical outcomes between two strategies of transfusion in oncologic surgery - liberal or restrictive

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer after major abdominal surgery requiring post-operative ICU admission
* Adults patients

Exclusion Criteria:

* Age less than 18 year
* Hematologic Malignances
* Intensive care unit permanence lower than 24 hours
* Renal Chronic Failure in Renal Replacement Therapy
* Karnofsky Status < 50
* Previous anemia (hemoglobin lower than 9 g/dL)
* Previous thrombocytopenia (platelet number lower than 50.000/mm3)
* Previous known coagulopathy
* Anticoagulation therapy
* Those unable to receive blood transfusion
* Patients who refused participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Composite end-point of mortality and severe complication | 30 days
  • The primary purpose of this study is to compare clinical outcomes after oncologic surgery in patients submitted to different strategies of red blood cell transfusion

SECONDARY OUTCOMES:
Hospital Length of Stay | 60 days
  • To compare length of stay in ICU, length of stay in Hospital, health-related quality of life and hospital costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836